CLINICAL TRIAL: NCT05294393
Title: Evaluation of Ropivacaine and Ropivacaine Plus Magnesium Sulphate Infiltration for Postoperative Analgesia in Patients Undergoing Thyroidectomy
Brief Title: Ropivacaine Plus Magnesium Sulphate Infiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Styliani Konstantinos Laskou, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3.468
Record Dates: First submitted 2022-03-01; First posted 2022-03-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Thyroid Diseases; Parathyroid Diseases; Postoperative Pain; Anesthesia, Local
Keywords: thyroidectomy; parathyroidectomy; local wound infiltration; ropivacaine; magnesium sulphate
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases; Pain, Postoperative | interventions — Ropivacaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N/S 0.9% (Placebo Comparator): Wound infiltration with 12 ml of N/S 0.9% at the end of surgery before wound closure
  Interventions: Drug: Placebo Comparator: N/S 0.9%
- Ropivacaine 10% (Active Comparator): Wound infiltration with 12 ml solution of 100mg ropivacaine at the end of surgery before wound closure
  Interventions: Drug: Ropivacaine 10%
- Ropivacaine 10% magnesium sulphate 10mg/kg (Experimental): Wound infiltration with 12 ml solution of 100mg ropivacaine plus magnesium sulphate 10mg/kg at the end of surgery before wound closure
  Interventions: Drug: Ropivacaine 10% plus magnesium sulphate 10mg/kg

INTERVENTIONS:
Drug: Placebo Comparator: N/S 0.9% — 12 ml N/S 0.9% at the end of surgery
  Arms: N/S 0.9%
Drug: Ropivacaine 10% — 12 ml solution of 100mg ropivacaine at the end of surgery
  Arms: Ropivacaine 10%
Drug: Ropivacaine 10% plus magnesium sulphate 10mg/kg — 12 ml solution of 100mg ropivacaine plus magnesium sulphate 10mg/kg at the end of surgery
  Arms: Ropivacaine 10% magnesium sulphate 10mg/kg

SUMMARY:
In the domain of endocrine gland surgery, thyroidectomy is the most common procedure. Patients report moderate to severe discomfort postoperatively, which is induced by a variety of mechanisms, the most common of which are cervical incision and surgical maneuvers. The other two causes are endotracheal intubation and neck overextension. Incisional pain, odynophagia, dysphagia, neck and shoulder pain have all been reported as sources of discomfort.However, it seems that this discomfort has a time limit, with a considerable decrease in pain scores that will last 24 to 36 hours. Pain is felt more profoundly within the first few hours after surgery, peaking at 6 hours, with patients requesting further analgesic medication.

Surgical wound infiltration can inhibit this procedure by preventing the alginate signal from reaching the incision site's receptors. According to the multimodal analgesia trends, magnesium sulfate can be added to the ropivacaine solution. Magnesium acts as an NMDA (N-methyl-D-aspartate) receptor antagonist, inhibiting cerebral sensitization to peripheral pain stimuli while reducing pre-existing hyperalgesia.

It becomes evident that this combination could contribute to attain the maximum analgesic efficacy. So, if any superiority of ropivacaine plus magnesium sulphate over ropivacaine could be demonstrated this would be very helpful in providing sufficient analgesic effects with a low incidence of adverse effects, while enhancing the option of one day surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Surgical indication for Total thyroidectomy
* Surgical indication forparathyroidectomy

Exclusion Criteria:

* Patients < 18 years old
* Prior neck operation
* Lateral neck dissection
* Patient with history of chronic opioid use
* Patient with chronic pain syndromes
* Patient with allergy to ropivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of Ropivacaine Plus Magnesium Sulphate Infiltration vs Ropivacaine | 24 postoperative hours
  Calculation of the total post-operative analgesic doses administered, converted to effective mg of morphine.

SECONDARY OUTCOMES:
Incisional Pain | 30 minutes ,1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours
  Incisional Pain will be measured by Visual Analogue Scale (VAS) pain questionnaire
Subjective measurements 1 | 30 minutes before the infiltration, 6 hours and 24 hours postoperatively
  Alterations in cortisol in μg/dl
Subjective measurements 2 | 30 minutes before the infiltration, 6 hours and 24 hours postoperatively
  Alterations in Tumor Necrosis Factor a (TNF-a) in pg/ml
Subjective measurements 3 | 30 minutes before the infiltration, 6 hours and 24 hours postoperatively
  Alterations in Interleukin 6 (IL-6) in pg/ml
Complications | 24 hours, 7 days
  Adverse effects of the infiltrated agents

CONTACTS AND LOCATIONS:
Overall Officials: Styliani K Laskou, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University, Thessaloniki, Other, Greece

IPD SHARING:
Plan to Share IPD: No